CLINICAL TRIAL: NCT00051181
Title: A Safety and Efficacy Study of Travoprost 0.004% Compared to Latanoprost 0.005% in Patients With Chronic Angle-Closure Glaucoma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-38
Record Dates: First submitted 2003-01-03; First posted 2003-01-07 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma, Angle-Closure; Ocular Hypertension
Keywords: Glaucoma; POAG; OAG; OHT
MeSH Terms: conditions — Glaucoma, Angle-Closure; Ocular Hypertension; Glaucoma | interventions — Travoprost; Latanoprost

INTERVENTIONS:
Drug: Travoprost (0.004%)
Drug: Latanoprost (0.005%)

SUMMARY:
To demonstrate that the intraocular pressure(IOP)-lowering efficacy of Travoprost (0.004%) is equal or better than that of Latanoprost 0.005% in patients with chronic angle-closure glaucoma.

ELIGIBILITY:
Adult patients of any race and either sex with chronic angle-closure glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Asia, Fort Worth, Texas, United States
- Australia, Sydney, Australia